CLINICAL TRIAL: NCT05278624
Title: Evaluation of the Safety and Efficacy of Topical Roflumilast Cream in the Treatment of Facial Papulopustular Rosacea
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dermatology Consulting Services, PLLC (Network)
Responsible Party: Principal Investigator, Zoe Diana Draelos, MD, President and Primary Investigator, Dermatology Consulting Services, PLLC
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DCS-41-20
Record Dates: First submitted 2022-03-04; First posted 2022-03-14 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Rosacea
MeSH Terms: conditions — Rosacea

STUDY DESIGN:
Intervention Model Description: Single site double blind vehicle controlled
Who Masked: Participant, Investigator
Masking Description: Identical tubes will be dispensed numerically with 50% containing vehicle and 50% containing vehicle plus active
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active plus vehicle arm (Active Comparator): Subjects will be dispensed a tube containing roflumilast and vehicle in topical formulation
  Interventions: Drug: Roflumilast Cream
- Vehicle arm (Placebo Comparator): Subjects will be dispensed a tube containing vehicle only in a topical formulation
  Interventions: Drug: Roflumilast Cream

INTERVENTIONS:
Drug: Roflumilast Cream — Topical Cream

SUMMARY:
This is a double blind single site vehicle controlled study. The following activities will be conducted at each visit.

Baseline Research Center Visit Obtain a signed and dated, written ICF prior to any study-related procedures.· Obtain demographic data· Assign subject number based on the order in which subjects present to the research center· Obtain medical/surgical history· Obtain concomitant medications· Assess eligibility based on inclusion/exclusion criteria· Collect blood and urine samples for clinical laboratory tests and send to the central laboratory· Perform serum pregnancy test in all women of child bearing potential (WOCBP)· Obtain vitals· Assess IGA, inflammation, erythema· Perform facial lesion counts· Perform local signs and symptoms assessments· Perform Columbia Suicide Severity Rating Scale (C-SSRS) for baseline visit· Randomize subject and dispense Investigational Study Medication and use instructions along with compliance diary· Schedule return visit

Week 2 Phone Call· Reassess medical/surgical history· Reassess concomitant medications· Assess adverse events· Assess compliance

Weeks 4, 8 Research Center Visit Reassess medical/surgical history· Reassess concomitant medications· Assess adverse events· Collect a urine sample from female subjects of childbearing potential for a urine pregnancy test· Obtain vitals· Assess IGA, inflammation, erythema· Perform facial lesion counts· Perform local signs and symptoms assessments· Perform Columbia Suicide Severity Rating Scale (C-SSRS) for return visits· Assess compliance diary and Investigational Study Medication, collect used Investigational Study Medication and redispense as necessary· Schedule return visit

Week 12 Research Center Visit· Reassess medical/surgical history· Reassess concomitant medications· Assess adverse events· Collect a urine sample from female subjects of childbearing potential for a urine pregnancy test· Collect blood and urine samples for clinical laboratory tests and send to the central laboratory· Obtain vitals· Assess IGA, inflammation, erythema· Perform facial lesion counts· Perform local signs and symptoms assessments· Perform Columbia Suicide Severity Rating Scale (C-SSRS) for return visits· Assess compliance diary and Investigational Study Medication· Collect diary and Investigational Study Medication· Release subject from study participation

ELIGIBILITY:
Inclusion Criteria:

1. Participants legally competent to sign and give informed consent or, in the case of adolescents, assent with consent of a parent(s) or legal guardian, as required by local laws.
2. Males and females ages 18 years to 70 years (inclusive) at the time of consent.
3. Clinical diagnosis of facial rosacea as confirmed by the investigator.
4. Subjects must have moderate to severe rosacea (as per IGA score) and at least 15 and not more than 75 inflammatory facial papules and pustules.
5. Subjects must have no more than 2 nodules on the face.
6. Subjects must have a definite clinical diagnosis of facial rosacea severity at least grade 3 as defined below:Score Grade Definition 0 Clear No inflammatory papules or pustules 1 Almost Clear Few inflammatory papules or pustules 2 Mild Several inflammatory papules or pustules 3 Moderate Moderate number of inflammatory papules or pustules and no nodules 4 Severe Many inflammatory papules or pustules, and up to 2 nodules Nodules will be reported separately and not included in the inflammatory lesion counts.
7. Subjects must have presence or history of erythema and/or flushing on the face.
8. Subjects willing to minimize external factors that might trigger rosacea flare-ups (eg, spicy, thermally hot foods and drinks, hot environments, prolonged sun exposure, strong winds, and alcoholic beverages).
9. Subjects who use make-up must have used the same brands/types of make-up for a minimum period of 14 days prior to study entry and must agree to not change make-up brand/type or frequency of use throughout the study.
10. Females of childbearing potential (FOCBP) must have a negative serum pregnancy test at Screening (Visit 1) and a negative urine pregnancy test at Baseline (Visit 2). In addition, sexually active FOCBP must agree to use at least one form of highly effective contraception throughout the trial. Highly effective forms of contraception include: oral/implant/injectable/transdermal contraceptives, intrauterine device, and partner's vasectomy. If barrier methods are used (e.g., condom with spermicide, diaphragm with spermicide), then 2 forms of conception are required in association with spermicide. The use of abstinence as a contraceptive measure is acceptable as long as this is a consistent part of a lifestyle choice and an acceptable backup method has been identified if the subject becomes sexually active.
11. Females of non-childbearing potential must either be pre-menarchal, or post-menopausal with spontaneous amenorrhea for at least 12 months (post-menopausal status should be confirmed with FSH testing) or have undergone surgical sterilization (permanent sterilization methods include hysterectomy, bilateral oophorectomy, hysteroscopic sterilization, bilateral tubal ligation or bilateral salpingectomy).
12. Subjects in good health as judged by the Investigator, based on medical history, physical examination, vital signs, serum chemistry labs, hematology values, and urinalysis.
13. Subjects are considered reliable and capable of adhering to the Protocol and visit schedule, according to the judgment of the Investigator.

Exclusion Criteria:

1. Subjects with any serious medical condition or clinically significant laboratory, vital signs, or physical examination abnormality that would prevent study participation or place the subject at significant risk, as judged by the Investigator
2. Subjects who cannot discontinue medications and treatments prior to the Baseline visit and during the study according to Excluded Medications and Treatments (Table 1).
3. Subjects who have unstable rosacea.
4. Presence of any skin condition on the face that would interfere with the diagnosis or assessment of rosacea.
5. Moderate or severe rhinophyma, dense telangiectasia or plaque-like facial edema.
6. Excessive facial hair (eg, beards, sideburns, moustaches, etc.) that would interfere with diagnosis or assessment of rosacea.
7. History of hypersensitivity or allergy to the study drug or of any other component of the formulation.
8. Severe erythema, dryness, scaling, pruritus, stinging/burning, or edema.
9. Active ocular rosacea (eg, conjunctivitis, blepharitis, or keratitis) of sufficient severity to require topical or systemic antibiotics.
10. Use within 6 months prior to Baseline of oral retinoids (eg, Accutane®) or therapeutic vitamin A supplements of greater than 10,000 units/day (multivitamins are allowed).
11. Initiation of use of estrogens or oral contraceptives less than 3 months prior to Baseline.
12. Use within 1 month prior to Baseline of:a. Topical retinoids to the face.b. Systemic antibiotics known to have an impact on the severity of facial rosaceac. Systemic corticosteroids (Note: intranasal and inhalation corticosteroids do not require a washout and maybe used throughout the trial if the subject is on a stable dose).
13. Use within 2 weeks prior to Baseline of:a. Topical corticosteroids.b. Topical antibiotics.c. Topical medications for rosacea.
14. Use of a sauna during the 2 weeks prior to Baseline and during the study.
15. Wax epilation of the face within 2 weeks prior to Baseline.
16. Consumption of excessive alcohol, abuse of licit or illicit drugs, or a condition that, in the opinion of the Investigator, could compromise the subject's ability to comply with study requirements.
17. Participation in activities that involve excessive or prolonged exposure to sunlight or weather extremes, such as wind or cold.
18. Presence of any clinically significant condition or situation, other than the condition being studied, that in the opinion of the Investigator would interfere with the study evaluations or optimal participation in the study.
19. Participation in an investigational drug study within 30 days prior to Baseline.
20. Prior laser therapy or phototherapy or other cosmetic procedures to the face that might affect rosacea in the opinion of the Investigator within 6 months of study entry.
21. Subjects who have received oral roflumilast or other PDE4 inhibitors (apremilast) within the past 4 weeks.
22. Subjects who have a history of or currently active depression, suicidal ideation, or suicidal tendencies as determined by verbal medical history.
23. Subjects with seborrheic dermatitis/rosacea overlap.
24. Subjects who are unwilling to refrain from using a tanning bed or other LEDs as well as outdoor tanning or excessive sun exposure for 4 weeks prior to Baseline and during the study.
25. Subject has a known or suspected allergy to Roflumilast cream or to excipients in Roflumilast cream (petrolatum, isopropyl palmitate, methylparaben, propylparaben, diethylene glycol monoethyl ether, hexylene glycol, cetylstearyl alcohol, dicetyl phosphase and ceteth-10 phosphate).
26. Subjects who have received oral roflumilast (Daxas®, Daliresp®) within the past 4 weeks.
27. Known or suspected: · severe renal insufficiency or moderate to severe hepatic disorders · history of chronic infectious disease (e.g., hepatitis B, hepatitis C, or human immunodeficiency virus (HIV)
28. Females who are pregnant, wishing to become pregnant during the study, or are breast-feeding.
29. Previous treatment with roflumilast cream.
30. Subjects with a history of chronic alcohol or drug abuse within 6 months of initiation of study Investigational Study Medication.
31. History of and/or concurrent condition of serious hypersensitivity (anaphylactic shock or anaphylactoid reaction) to PDE-4 inhibitors.
32. Current or a history of cancer within 5 years with the exception of fully treated skin basal cell carcinoma, cutaneous squamous cell carcinoma or carcinoma in situ of the cervix.
33. Subjects with a history of a major surgery within 8 weeks prior to Baseline or has a major surgery planned during the study.
34. Subjects who are unable to communicate, read or understand the local language, or who display another condition, which in the Investigator's opinion, makes them unsuitable for clinical study participation.
35. Subjects that are family members of the clinical study site, clinical study staff, or Arcutis, or family members of enrolled subjects.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-04-15 (Actual); Primary Completion 2023-02-17 (Actual); Study Completion 2023-02-17 (Actual)

PRIMARY OUTCOMES:
Primary Outcome Measure | 12 Weeks
  The primary outcome measure is the reduction in rosacea facial inflammatory lesion count from baseline as compared to week 12.

SECONDARY OUTCOMES:
Secondary Outcome Measure | 12 weeks
  The secondary outcome measure is the percent change in the rosacea Investigator Global Assessment (IGA) from baseline as compared to week 12.

CONTACTS AND LOCATIONS:
Locations (1):
- Dermatology Consulting Services, PLLC, High Point, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
No data will be shared from this pilot study.